CLINICAL TRIAL: NCT00596934
Title: Nonalcoholic Steatohepatitis: is Leptin an Etiological Factor (Phase 2).
Brief Title: Recombinant Leptin Therapy for Treatment of Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elif Oral (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Elif Oral, Associate Prof of Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R03DK074488 (NIH); R03DK074488 (NIH); Protocol 2145 (MCRU); Amylin Protocol 20050119; DRDA 643938K3
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Fatty Liver Disease, Nonalcoholic
Keywords: Nonalcoholic fatty liver disease; Insulin resistance; Obesity; Leptin therapy; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Obesity | interventions — metreleptin; recombinant methionyl human leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metreleptin treatment group (Experimental): Treatment group
  Interventions: Drug: metreleptin

INTERVENTIONS:
Drug: metreleptin — 0.1 mg/kg/day once a day via subcutaneous injections
  Other Names: (originally A100, recombinant-human-Methionyl-leptin

SUMMARY:
Nonalcoholic steatohepatitis (or NASH) is known to be caused by deposition of fat in the liver and development of scarring. This condition occurs more frequently in overweight and obese persons. It is often associated with resistance to the actions of insulin hormone. Fat cells secrete a hormone called leptin. Recently, we have learned that obese or overweight persons make too much leptin, which may contribute to insulin resistance. Paradoxically, patients who do not have any fat cells, also have insulin resistance. In these patients, insulin resistance is caused by the absence of leptin and leptin replacement significantly improves insulin resistance and fat deposition in the liver. In an earlier study, we determined the leptin levels in patients with NASH and how these levels are related to body fat levels as well as responsiveness to insulin. We saw that a subgroup of patients with NASH have relatively low levels of leptin in contrast to the amount of body fat they had. We now would like to see if restoring leptin levels to normal will improve the disease process in these patients. Our study patients will be male patients, aged between 18 and 65 (inclusive), who do not have any other cause for their liver disease. We have put some restrictions in body size such that a spectrum of patients from normal weight to obese range would be included. They will also demonstrate low leptin levels (levels similar to only 25% of normal population). We will use a genetically engineered form of leptin manufactured by Amylin Inc. given via injections under the skin. We plan to continue therapy for a period of one year and evaluate the change in liver disease by a liver biopsy. We will also follow the metabolic parameters and body composition characteristics that we examined in our earlier study. We expect that patients with low blood leptin levels will show improvement in their liver disease and insulin resistance when their blood leptin levels are restored to normal.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NASH
* Circulating fasting leptin <9 ng/mL (staggered criteria for different BMI levels)

Exclusion Criteria:

* Presence of advanced liver disease (as evidenced by abnormal synthetic function, abnormal prothrombin time or albumin)
* Presence of clinical lipodystrophy
* Presence of other liver disease
* Presence of clinical diabetes (fasting >126 mg/dL or 2 hour post 75 g-glucose >200 mg/dL or random glucose >200 mg/dL with presence of diabetes symptoms or known history of diabetes)
* Any medication for treatment of NASH or obesity
* Presence of HIV
* Inability to give informed consent
* Presence of end-stage renal disease, any type of active cancer, or >class 2 congestive heart failure ((New York Heart Association Functional Classification System), based on medical history and physical examination
* Presence of any other condition that limits life expectancy to <2 years
* Active infection (may be transient)
* Any other condition in the opinion of the investigators that may impede successful data collection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akinci B, Subauste A, Ajluni N, Esfandiari NH, Meral R, Neidert AH, Eraslan A, Hench R, Rus D, McKenna B, Hussain HK, Chenevert TL, Tayeh MK, Rupani AR, Innis JW, Mantzoros CS, Conjeevaram HS, Burant CL, Oral EA. Metreleptin therapy for nonalcoholic steatohepatitis: Open-label therapy interventions in two different clinical settings. Med. 2021 Jul 9;2(7):814-835. doi: 10.1016/j.medj.2021.04.001. Epub 2021 May 12. PMID 35291351
- See also: PIs Web site — http://www.uofmhealth.org/profile/83/elif-oral-md

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from February 2007 and concluded in October 2007.
Pre-assignment Details: One of ten enrolled participants screen failed during baseline visit, liver biopsy showed no non-alcoholic steatohepatitis. Therefore he is not included in any tables or analyses.
Groups:
- NASH02: Treatment group
  metreleptin : 0.1 mg/kg/day once a day via subcutaneous injections
Period: Overall Study
Arm/Group | NASH02
Started | 9
Completed | 7
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Metreleptin Treatment Arm: Treatment group
  metreleptin : 0.1 mg/kg/day once a day via subcutaneous injections
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 44.3 [32 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9
Non-alcoholic steatohepatitis (NASH) score [Mean (Standard Deviation); unit: units on a scale] — NASH scale: 0 - 14. The higher the NASH score the more severe the liver disease.
  units on a scale | 8.1 (3.3)
Body Weight [Mean (Standard Deviation); unit: kg] | 90.9 (9.0)
Liver fat percentage by Magnetic Resonance Imaging (MRI - Dixon method) [Mean (Standard Deviation); unit: liver fat percentage] — For determination of hepatic fat content by MRI and MR spectroscopy in patients, a series of out-phase and in-phase MRI at multiple flip angles are used. By combination of out-phase and in-phase MRI at multiple flip-angles and TE times, relaxation-time effects can be removed to yield quantitative intra-hepatic (and other organs') fractional fat content throughout the liver in a few breath-hold intervals.
  liver fat percentage | 19.0 (7.7)
Liver function test: Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] — Normal range for laboratory values: <=35 IU/L
  IU/L | 50.9 (19.4)
Liver function test: Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: IU/L] — Normal range for laboratory values: 8 - 30 IU/L
  IU/L | 33.5 (13.3)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] — Normal range for laboratory values: 73 - 100 mg/dL
  mg/dL | 98.1 (7.2)
Insulin Resistance: homeostatic model assessment (HOMA) [Mean (Standard Deviation); unit: mU/L x mg/dL] — HOMA values are based on fasting insulin and glucose concentrations and calculated as fasting insulin concentration (mU/L) x fasting glucose concentration (mg/dL)/405
  mU/L x mg/dL | 7.4 (3.2)
Fasting triglycerides [Mean (Standard Deviation); unit: mg/dL] — Normal range for laboratory values: <150 mg/dL
  mg/dL | 129.4 (66.2)

OUTCOME MEASURES:

1. Primary Outcome: Non-alcoholic Steatohepatitis Score as Determined by Liver Histopathology at 12 Months
Description: Non-alcoholic steatohepatitis (NASH) score after approximately one year of treatment with metreleptin. Total NASH scores can range from 0 to 14. The higher the NASH score the more severe the liver disease.
Time Frame: 1 year
Population: Individuals who completed the year of metreleptin treatment and had follow-up liver biopsies after one year.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
units on a scale | 5 (1.73)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Differences in each collected parameter will be evaluated using a paired t-test. If data are skewed such as in triglyceride levels, nonparametric tests will be used. P<0.05 will be considered significant. If a significant difference can be demonstrated between baseline and 1-year results, a large scale, placebo-controlled trial will be designed using the data obtained from this pilot study; Test type: Superiority or Other; p = 0.015, t-test, 2 sided

2. Secondary Outcome: Body Weight at 12 Months
Description: Body weight (kg) after one year of treatment on metreleptin for patients that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: Subjects that completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Metreleptin Treatment Arm: Treatment group
  metreleptin: 0.1 mg/kg/day once a day via subcutaneous injections
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
kg | 86.4 (9.9)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Liver Fat Percentage by Magnetic Resonance Imaging (MRI - Dixon Method) at 12 Months
Description: For determination of hepatic fat content by MRI and MR spectroscopy in patients, a series of out-phase and in-phase MRI at multiple flip angles are used. By combination of out-phase and in-phase MRI at multiple flip-angles and TE times, relaxation-time effects can be removed to yield quantitative intra-hepatic (and other organs') fractional fat content throughout the liver in a few breath-hold intervals.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: liver fat percentage
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
liver fat percentage | 13.7 (9.1)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p = 0.074, t-test, 2 sided — p = 0.074

4. Secondary Outcome: Liver Function Test: Alanine Aminotransferase (ALT) Values at 12 Months
Description: ALT value in subjects that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: 7 subjects who completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
IU/L | 44.3 (29.1)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

5. Secondary Outcome: Liver Function Test: Aspartate Aminotransferase (AST) Values at 12 Months
Description: AST value in subjects that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: 7 subjects who completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Metreleptin Treatment Group
Number analyzed (Participants) | 7
IU/L | 34.9 (13.9)
Statistical Analysis 1: Comparison: Metreleptin Treatment Group; Test type: Superiority or Other; p = 0.006, t-test, 2 sided

6. Secondary Outcome: Fasting Glucose Value at 12 Months
Description: Fasting glucose value in subjects that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: 7 subjects who completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
mg/dL | 92.1 (5.9)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p = 0.023, t-test, 2 sided

7. Secondary Outcome: Fasting Triglycerides Value at 12 Months
Description: Fasting triglyceride value in subjects that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: 7 subjects who completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
mg/dL | 146.4 (75.7)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p = 0.195, t-test, 2 sided — p-value = 0.195

8. Secondary Outcome: Insulin Resistance: Homeostatic Model Assessment (HOMA) at 12 Months
Description: HOMA values in subjects that completed 12 months of metreleptin treatment.
Time Frame: 1 year
Population: 7 subjects who completed 12 months of metreleptin treatment.
Measure: Mean (Standard Deviation); unit: mU/L x mg/dL
Arm/Group | Metreleptin Treatment Arm
Number analyzed (Participants) | 7
mU/L x mg/dL | 4.1 (3.0)
Statistical Analysis 1: Comparison: Metreleptin Treatment Arm; Test type: Superiority or Other; p = 0.026, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 13 months from patient baseline appointment.
Description: Adverse event data collected from patient's baseline study appointment till one month following patient's 12 month study appointment.
Arm/Group | Metreleptin Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin Treatment Arm (N=9)
toxoplasmosis (Blood and lymphatic system disorders) | 1 (1) — add description of advent.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin Treatment Arm (N=9)
left side muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
vertigo (Nervous system disorders) | 1 (1)
polyuria (Renal and urinary disorders) | 1 (1)
actinic keratoses (Skin and subcutaneous tissue disorders) | 1 (10)
haematuria (Renal and urinary disorders) | 1 (1)
rectal pressure with ejaculation (Reproductive system and breast disorders) | 1 (1)
right sternocleidomastoid lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
right axilla lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a non-blinded, non-placebo controlled proof of concept trial. Out of the 9 patients, there were 7 completers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No